CLINICAL TRIAL: NCT02740803
Title: Total Salivary Fluoride Concentration of Healthy Adult Subjects Following Toothbrushing With Different Formulations of Fluoridated Toothpastes With and Without Post-brushing Water Rinsing. A Double Blinded Randomised Controlled Trial
Brief Title: Total Salivary Fluoride Concentration of Healthy Adult Subjects Following Toothbrushing With Different Formulations of Fluoridated Toothpastes With and Without Post-brushing Water Rinsing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Marwah Albahrani, Post-graduate Professional Doctorate of Paediatric Dentistry, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16/YH/0015
Record Dates: First submitted 2016-02-24; First posted 2016-04-15 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- NaF - R (Experimental): Participants will use sodium fluoride toothpaste (1,450 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: Sodium fluoride toothpaste 1,450 ppmF
- NaF - NR (Experimental): Participants will use sodium fluoride toothpaste (1,450 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: Sodium fluoride toothpaste 1,450 ppmF
- NaMFP- R (Experimental): Participants will use sodium monofluorophosphate toothpaste (1,450 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: sodium monofluorophosphate toothpaste 1,450 ppmF
- NaMFP- NR (Experimental): Participants will use sodium monofluorophosphate toothpaste (1,450 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: sodium monofluorophosphate toothpaste 1,450 ppmF
- SnF + NaF - R (Experimental): Participants will use stannous fluoride combined with sodium fluoride toothpaste (1,450 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: stannous fluoride combined with sodium fluoride toothpaste 1,450 ppmF
- SnF + NaF - NR (Experimental): Participants will use stannous fluoride combined with sodium fluoride toothpaste (1,450 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: stannous fluoride combined with sodium fluoride toothpaste 1,450 ppmF
- NaF + NaMFP - R (Experimental): Participants will use sodium fluoride combined sodium monofluorophosphate toothpaste (1,450 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: sodium fluoride combined sodium monofluorophosphate toothpaste 1,450 ppmF
- NaF + NaMFP - NR (Experimental): Participants will use sodium fluoride combined sodium monofluorophosphate toothpaste (1,450 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: sodium fluoride combined sodium monofluorophosphate toothpaste 1,450 ppmF
- AmF - R (Experimental): Participants will use amine fluoride toothpaste (1,400 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: Amine fluoride toothpaste 1,400 ppmF
- AmF - NR (Experimental): Participants will use amine fluoride toothpaste (1,400 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: Amine fluoride toothpaste 1,400 ppmF
- 0 Fluoride - R (Experimental): Participants will use non-fluoridated toothpaste (0 ppmF) to brush for two minutes followed by rinsing with distilled water.
  Interventions: Other: Non-fluoridated toothpaste 0 ppmF
- 0 Fluoride - NR (Experimental): Participants will use non-fluoridated toothpaste (0 ppmF) to brush for two minutes not followed by rinsing with distilled water.
  Interventions: Other: Non-fluoridated toothpaste 0 ppmF

INTERVENTIONS:
Other: Sodium fluoride toothpaste 1,450 ppmF
  Arms: NaF - NR; NaF - R
Other: sodium monofluorophosphate toothpaste 1,450 ppmF
  Arms: NaMFP- NR; NaMFP- R
Other: stannous fluoride combined with sodium fluoride toothpaste 1,450 ppmF
  Arms: SnF + NaF - NR; SnF + NaF - R
Other: sodium fluoride combined sodium monofluorophosphate toothpaste 1,450 ppmF
  Arms: NaF + NaMFP - NR; NaF + NaMFP - R
Other: Amine fluoride toothpaste 1,400 ppmF
  Arms: AmF - NR; AmF - R
Other: Non-fluoridated toothpaste 0 ppmF
  Arms: 0 Fluoride - NR; 0 Fluoride - R

SUMMARY:
Caries prevalence has declined significantly since the introduction of fluoridated toothpastes. Since then, different toothpaste formulations and concentrations have been introduced to the market with varying levels of efficacy. There are several commercially available toothpastes to choose from and only with the aid of sound methodological research, can the best evidence-based oral education advice be delivered.

This is a double-blinded randomised controlled trial that aims to measure the salivary fluoride concentration following tooth-brushing with several toothpaste formulations. Power calculations were performed using PASS 11.0 software, and calculations showed that 3 participants are needed in each group in order for results to be considered as significant. We will aim to recruit five to seven participants in each of the 12 groups. Research will be publicised by means of flyers and circulating emails amongst University of Leeds students. Information sheets will be provided to all participants and informed consent will be obtained.

Each participant will brush with one of 6 different formulations of toothpastes either with or without water rinsing post-brushing. Participants will randomly be assigned to groups using an online random team generator. Saliva will be collected six times once before brushing and at 1, 15, 30, 60 and 90 minutes post-brushing. Samples will be analysed using fluoride ion-specific sensitive electrode connected to an ion analyser.

A statistician's help will be sought for analysis of the results. After the analysis stage, the codes of the toothpastes will be broken.

DETAILED DESCRIPTION:
Study design:

Double-Blinded Randomised controlled trial

Study aim:

This is an in vivo study that aims to compare the salivary fluoride concentrations of different fluoride formulations in the form of toothpaste with and without post-brushing water rinsing.

Study objectives:

To compare the salivary fluoride concentrations of different fluoride formulations in the form of toothpaste, with and without post-brushing water rinsing. Toothpaste formulations are to include: sodium fluoride (NaF), sodium monofluorophosphate (MFP), sodium fluoride plus sodium monofluorophosphate combined (NaF + MFP), Amine fluoride (AmF) and stannous fluoride and sodium fluoride combined (SnF + NaF). Fluoride-free toothpaste will serve as a control in this study. Concentration is to be standardised for all the formulations.

Results of this study would reflect on the oral hygiene instructions given to patients in term of tooth brushing frequency, fluoride-containing dentifrices of different formulations and post-brushing rinsing practice.

Null hypothesis:

The null hypotheses for this study are:

All of the following toothpaste formulations have no significant difference in term of salivary clearance rate:

oNon-fluoridated toothpaste oSodium fluoride (Naf) toothpaste oSodium fluoride and sodium monofluorophosphate combined toothpaste (NaF+ MFP) oStannous fluoride and sodium fluoride combined (SnF+NaF) toothpaste oAmine fluoride toothpaste (AmF) oSodium monofluorophosphate toothpaste

Materials under investigation:

The experimental materials to be investigated are taken from the list of the available brands in UK published in delivering better oral health: an evidence-based toolkit for prevention.

* Control toothpaste (0 ppmF)
* Sodium fluoride toothpaste 1,450 ppm F
* Sodium monofluorophosphate toothpaste1,450 ppm F
* Sodium monofluorophosphate + sodium fluoride combined toothpaste 1,450 ppm F
* Stannous fluoride + sodium fluoride combined toothpaste1,450 ppm F
* Amine fluoride toothpaste 1,400 ppm F

Sample size and power calculation:

Statistical advice was sought and sample size calculation was performed using PASS 11.0 software. A sample of at least 3 participants is needed for each group. The study aims to test 12 different groups, with 5 participants in each group, giving a total number of 60 participants.

As recommended by the Research Ethics Committee (REC) committee the investigators have rerun the power calculations again, using raw data from Issa and Toumba, 2004 without the data from the control groups, and similar results were obtained.

The Research Ethics Committee (REC) has approved increasing the sample size to at least 120 participants in total.

Obtaining informed consent Contact details are enclosed in the recruitment emails, flyers and information sheet. Information sheet and a copy of the consent sheet will be sent to participants by emails, post or they can come and pick it up at their comfort. Participants will still have the opportunity to contact the lead researcher for further questions or queries through either her contact number or her university email.

The information sheet to this research study will be used as an invitation letter as well.

On the research day, consent sheets will be explained and an informed consent will be obtained from all participants. The original copy of the consent sheet will be kept by the lead researcher and participants will retain the copy of their signed consent form.

Anonymising patients Participants will be identified by a numerical number rather than their names.

Blinding toothpaste groups A third party will put toothpastes in small identical containers labelled with the group number (G1-12), batch number and expiry date. This will be done randomly using the following website.

https://www.randomlists.com/team-generator A file will be attached in the checklist explaining the randomisation process.

Random assignments of toothpastes to participants With aid of the following website (https://www.randomlists.com/team-generator), each reference number (participant number) will be randomly assigned to one of 12 groups.

Ethical approval:

All the required information will be provided to the Ethical committee (Leeds Health Authority / United Leeds Teaching Hospitals) in advance for ethical approval to be obtained prior commencement of the study.

Elective assessment of participants:

When participants contact the lead examiner (responding to the email or posters) about participating in the research study, volunteers will be asked several questions about their medical history (medical questionnaire) to determine whether they fall within ASA I and ASA II categories. Other ASA categories (ASA III or higher) will be excluded from the study, informed consent will not be obtained and no further information (i.e. information sheet) will be sent out.

If participants contact the lead examiner by email, then the medical history questionnaire will be asked by replying to their email. If however, the participants show interest over the phone, then the medical questionnaire will be obtained over the phone. For participants who show interest over the phone, they will be given the option whether they want the information sheet mailed to them, emailed or if they prefer to pick it up at their convenience.

For participants who are included in the research gender, age and carious status will be recorded on the assessment sheet. This information will remain anonymous and will not identify participants since each participant will be identified by a number.

After result analysis, results will be disseminated to all participants attached with an appreciation letter.

The American Society of Anaesthesiologist (ASA) Physical Status Classification ASA 1 A normal healthy patient ASA 2 A patient with mild systemic disease ASA 3 A patient with severe systemic disease ASA 4 A patient with severe systemic disease that is a constant threat to life ASA 5 A moribund patient who is not to survive without the operation ASA 6 A declared brained-dead patient whose organs are being removed for donor purposes

Publicity and recruitment of participants Participant recruitment will be performed by the means of recruitment flyers and circular emails. Recruitment flyers will be posted across the Worsley building of the University of Leeds (Level 6 and Level 7, Worsley building, West Yorkshire, LS2 9JT) and Leeds Dental Institute (Leeds, West Yorkshire, LS2 9LU). Circular emails will be emailed to all University students, after permission from the school's office. This means that the population targeted would be staff and students of the University of Leeds and possibly their families, visitors to the University of Leeds and patients under the care of Leeds Dental Institute.

The recruitment of NHS patients will follow a similar process to the other volunteers. Recruitment leaflets will be put at the reception and waiting areas of each different department. A copy of the information sheet and the consent sheet can be obtained from the receptionists upon request. Participants who wish to take part in this study will have to contact the lead examiner (Marwah Albahrani) through the contact details on the recruitment flyers and the information sheets. Informed consent will obtained following the procedure explained under the subheading "obtaining informed consent".

The emails will be short and the subject line will include a short description of the study followed by the word "circular". Subject line: Participant needed for tooth-brushing - Circular.

The email will start with:

'Circular email for use for recruitment of participants for study ref: Ethics reference number, approved by [INSERT NAME OF ETHICS SUBCOMMITTEE/PANEL].

This project contributes to the University's role in conducting research, and teaching research methods. You are under no obligation to reply to this email, however if you choose to, participation in this research is voluntary and you may withdraw at anytime. Please see attached for more details.

A copy of the recruitment flyer, the information sheet and consent sheet will be attached to the circular email.

Sending out appointments for participants An appointment message will be sent out to participant's contact numbers informing them with the date of the research appointment.

Message reminders one day before appointment A reminder message will be sent one day before the appointment. This will also include fasting and tooth-brushing instructions.

A list of which patient is going to be in which group will be published before the day of the appointment according to the blinding and randomisation procedures explained above.

For each participant, 1.0 ml whole mixed saliva will be collected in a plastic beaker labelled with their reference number, group, rinsing method and time interval. Participants will then be asked to brush their teeth with pre-weighed amount of toothpaste for 2 full minutes.

Depending on which group, participants will be either asked to spit the excess toothpaste and not rinse their mouth for the entire appointment or participants might be ask to rinse their mouth with 10 ml of water for 5 seconds.

Each participant will have a slip stating times at which their saliva samples (1.0 ml) will be collected. After each sample collection, the time interval will be ticked off on the slip. Participants will be waiting in the waiting room and will be instructed to refrain from eating or drinking during the length of their appointment. Saliva samples will be collected by the lead investigator (M. Albahrani) 6 times at the following time intervals: 0,1, 15, 30, 60 and 90 minutes.

Participants will be given £10 to compensate for their time, transport and food expenses.

Sample analysis Fluoride concentration will be measured using an ion-specific sensitive electrode connected to an ion analyser.

REPRODUCIBILITY OF THE MEASRUMENTS Reproducibility of the results will be checked by using fluoride ion standard solutions.

Data management and analysis

Two way mirroring ANOVA meaning that:

1. ANOVA statistical test will be performed comparing salivary fluoride concentration between the different time intervals of the same group.
2. ANOVA statistical test will be also performed to compare salivary fluoride concentration between different groups at the same time interval.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study should be ASA* I and ASA* II adult volunteers.
* Salivary flow rate of 0.1 ml / minute or more.
* Caries-free and non-caries free are to be included.

  * ASA stands for American society of Anesthesiologists grading system

Exclusion Criteria:

* Edentulous patients.
* Participants who are ASA* III or higher will be excluded.
* Allergy to any of the materials used in the study.
* Participants with orthodontic devices / braces.
* Participants with salivary flow rate of or below 0.1 ml / minute.
* Participants who are incapable of fasting for 4 hours.
* Participants who refuse to use fluoride-free toothpaste, or those who would want to have control over which toothpaste to use.
* Participants who cannot retain toothpaste and have to rinse after tooth brushing (ie. gagging due to toothpaste taste).

  * ASA stands for American society of Anesthesiologists grading system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Salivary fluoride concentration following brushing with different toothpaste formulations. | 0 minutes
  Prior brushing
Salivary fluoride concentration following brushing with different toothpaste formulations. | 1 minutes
  1 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations. | 15 minutes
  15 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations. | 30 minutes
  30 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations. | 60 minutes
  60 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations. | 90 minutes
  90 minutes postbrushing

SECONDARY OUTCOMES:
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 0 minutes
  Prior brushing
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 1 minutes
  1 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 15 minutes
  15 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 30 minutes
  30 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 60 minutes
  60 minutes postbrushing
Salivary fluoride concentration following brushing with different toothpaste formulations - with and without water rinsing | 90 minutes
  90 minutes postbrushing

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Dental Institute, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants will be informed that data will be anonymised so that they cannot be identified even in case of results dissemination (i.e peer-reviewed journals.
  Age, gender, sex, salivary rate per minutes, fluoride ion concentrations in saliva prior to brushing and post-brushing at 1, 15, 30, 60 and 90 minutes.

REFERENCES:
- [Derived] Albahrani MM, Alyahya A, Qudeimat MA, Toumba KJ. Salivary fluoride concentration following toothbrushing with and without rinsing: a randomised controlled trial. BMC Oral Health. 2022 Mar 3;22(1):53. doi: 10.1186/s12903-022-02086-5. PMID 35241051